CLINICAL TRIAL: NCT02148055
Title: Comparative Evaluation of IRM and Autopsy in the Evaluation of Intra Uterine Fetal Death.
Acronym: COMPER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of recruitment
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012/169/HP
Record Dates: First submitted 2014-05-22; First posted 2014-05-28 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Spontaneous Intra Uterine Fetal Death
Keywords: spontaneous intrauterine death; fetal MRI; autopsy
MeSH Terms: interventions — Autopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A group of 20 pregnant patients. (Other): 20 patients referred for intrauterine spontaneous fetal death explored by MRI and autopsy.
  Interventions: Other: Comparaison between MR and autopsy in the macroscopic evaluation of intra uterine death.

INTERVENTIONS:
Other: Comparaison between MR and autopsy in the macroscopic evaluation of intra uterine death.

SUMMARY:
Fetal intra uterine death is a rare event (incidence 2/1000 births) , unexpected and psychologically painful for the couple and the healthcare team. In this difficult context, it is essential to understand the etiology of death to guide the management of subsequent pregnancies. Among the investigations, foetopathologic examination is essential, but the examination of the brain is not possible in more than half of the cases due to the cerebral maceration due to the incompressible delay between death and expulsion.

The use of MRI as a diagnostic tool fetal post- mortem " virtual autopsy " performed before expulsion of the fetus is interesting because it would permit to obtain a macroscopic examination of the fetal brain, archivable, and a gain concerning the diagnosis. Thus, a normal MRI will exclude cerebral anatomical abnormality , stroke or bleeding . If MRI abnormalities are found , it will not only guide the foetopathologic review, but mainly to guide the etiology . On the other hand , it is a non-invasive tool and acceptability by the couple would be better than autopsy which is often refused by the couple in this difficult psychological context.

In this study , MRI will be given in addition to conventional autopsy in the painful waiting time between the time of diagnosis of death and expulsion without delaying care . If this study is validated , MRI may be systematically proposed in this indication or alternative to autopsy when it will be refused by the parents.

ELIGIBILITY:
Inclusion Criteria:

* Patient for which he was diagnosed with intra uterine death confirmed by ultrasound
* Mono fetal pregnancy,
* Term: 24 to 42 weeks' gestation
* Age> 18 years
* Patient having readen the letter of information and signed the consent.

Exclusion Criteria:

* Contraindication to MRI (heart valve, pacemaker, neurosurgical clips, claustrophobia, intraocular metallic foreign bodies)
* Maternal complications: bleeding during, eclampsia, placental hematoma retro, imminent work
* Twin pregnancy
* Patient under guardianship or trusteeship
* Patient not speaking and writing French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Recognition of anatomic cerebral structures evaluated by a common grid. | Before H 24 for MR. Bedore day 5 for autopsy.

SECONDARY OUTCOMES:
Recognition and mesurement of anatomic thoracic and abdominal structures by a common grid. | Before H24 for MR. Before day 5 for autopsy.
Recognition and mesurement of the placenta and umbilical cord. | Before H24 for IRM. Before day 5 for autopsy.
Comparaison of quality criteria of both exams. | Before H24 for MRI. Before day 5 for autopsy.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Hopitaux de Rouen, Rouen, France